CLINICAL TRIAL: NCT02463006
Title: Comparative Evaluation of Porous and Non Porous Variants of Bioactive Glass in the Treatment of Periodontal Intrabony Defects: A Cone Beam Computed Tomography Analysis
Brief Title: Porous and Non-porous Bone Grafts in Intra-bony Periodontal Defects
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Dr. D. Y. Patil Dental College & Hospital (Other)
Responsible Party: Principal Investigator, D. Gopalakrishnan, Professor, Dr. D. Y. Patil Dental College & Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DYPDCH/12/PG16
Record Dates: First submitted 2015-05-29; First posted 2015-06-04 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Periodontal Disease
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- porous bone graft group (Experimental): Intervention: Flap surgery procedure with porous bone grafting (Periooglass)
  Interventions: Drug: Porous variant of Bioactive Glass.
- Non-porous bone gaft group (Active Comparator): Intervention: Flap surgery procedure with non-porous bone grafting (Novabone morsels)
  Interventions: Drug: Non porous variant of Bioactive Glass.

INTERVENTIONS:
Drug: Porous variant of Bioactive Glass. — Flap surgery with Porous variant of Bioactive Glass.
  Arms: porous bone graft group
Drug: Non porous variant of Bioactive Glass. — Flap surgery with non-Porous variant of Bioactive Glass.
  Arms: Non-porous bone gaft group

SUMMARY:
Till date, no study has been reported in the literature where porous bioactive glass was used for the management of periodontal osseous defects. In this context, the present study is designed to assess the efficacy of the porous variant of bioactive glass and compare with that of nonporous variant using cone beam computed tomography.

DETAILED DESCRIPTION:
OBJECTIVES:

1. To evaluate clinically the periodontal healing with Porous variant of Bioactive Glass placed in the intra bony defects at an interval of 6 months.
2. To evaluate clinically the periodontal healing with Non Porous variant of Bioactive Glass placed in the intra bony defects at an interval of 6 months.
3. To evaluate the radiographic changes in the intra bony defect grafted with Porous variant of Bioactive Glass at baseline and an interval of 6 months.
4. To evaluate the radiographic changes in the intra bony defect grafted with Non Porous variant of Bioactive Glass at baseline and an interval of 6 months.
5. To compare clinically soft tissue healing for sites grafted with Porous variant of Bioactive Glass and sites grafted with Non Porous variant of Bioactive Glass in the treatment of periodontal intra bony defects at an interval of 6 months.
6. To compare the radiographic changes for sites grafted with Porous variant and sites grafted with Non Porous of Bioactive Glass in the treatment of periodontal intra bony defects at an interval of 6 months.

ELIGIBILITY:
Inclusion Criteria:

* INCLUSION CRITERIA

  1. Age: 18-55 years.
  2. Probing Depth >5mm.

Exclusion Criteria:

* EXCLUSION CRITERIA

  1. History of periodontal treatment last six months.
  2. Bleeding disorders.
  3. Gross oral pathology.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2014-01; Primary Completion 2014-09 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Change in relative attachment loss | 6 months

SECONDARY OUTCOMES:
Change in probing depth | 6 months
Change in plaque index | 6 months

REFERENCES:
- [Result] Gokhale ST, Dwarakanath CD. The use of a natural osteoconductive porous bone mineral (Bio-Oss) in infrabony periodontal defects. J Indian Soc Periodontol. 2012 Apr;16(2):247-52. doi: 10.4103/0972-124X.99270. PMID 23055593
- [Result] Wohlfahrt JC, Aass AM, Ronold HJ, Heijl L, Haugen HJ, Lyngstadaas SP. Microcomputed tomographic and histologic analysis of animal experimental degree II furcation defects treated with porous titanium granules or deproteinized bovine bone. J Periodontol. 2012 Feb;83(2):211-21. doi: 10.1902/jop.2011.110128. Epub 2011 Jun 21. PMID 21692628